CLINICAL TRIAL: NCT05949528
Title: Assessing Chronic Consciousness Disorders in Patients Using Clinical Evaluation With Resting-state EEG and ERPs: an Extensive Study Exploring Efficacy and Diagnostic Potential of EEG and ERP Measurements
Brief Title: Clinical Evaluation of Chronic Consciousness Disorders Using Resting-state EEG and ERP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: EEG assessment
Record Dates: First submitted 2022-03-14; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2022-10

CONDITIONS: Disorders of Consciousness
Keywords: resting-state electroencephalograms; ERP; microstate
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Electroencephalogram (EEG) refers to the resting state and event-related potential (ERP) of the brain.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Healthy controls (HCs): Healthy controls (HCs)
  Interventions: Other: no intervention
- Emerged from Minimally Conscious State (EMCS): Emerged from Minimally Conscious State (EMCS): recovery of functional object uses or communication from chronic
  Interventions: Other: no intervention
- Minimally conscious state (MCS): Minimally conscious state (MCS): have reproducible signs of awareness and exhibit fluctuations in consciousness
  Interventions: Other: no intervention
- Vegetative state (VS): Vegetative state (VS): can open their eyes and preserve sleep-wake cycles, but unaware of themselves and their surroundings
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Currently, there are significant challenges in the clinical assessment of patients with consciousness disorders, such as distinguishing between vegetative state (VS) and minimally conscious state (MCS), and predicting patient prognosis. This study aims to utilize different research techniques, such as auditory stimulation, as well as modified microstate methods, to enhance the disease classification and prognosis prediction of patients with chronic consciousness disorders.

DETAILED DESCRIPTION:
The investigators collected resting-state electroencephalograms (EEGs) and EEGs under various event-related potential (ERP) stimuli from patients with chronic consciousness disorders, and performed analyses on these data. The resting-state EEGs were subjected to spectral analysis and microstate analysis. The ERP EEGs were analyzed in the time domain, as well as for phase coupling and other measures.Using these computed indicators, the investigators use machine learning, deep learning, and other methods to predict disease classification and prognosis assessment in patients with chronic consciousness disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with COMA /VS/MCS
2. The course of disease was more than 4 weeks
3. The vital signs were stable and able to tolerate the test process
4. Complete skull
5. Right-handed, no history of ear disease or hearing loss before onset

Exclusion Criteria:

1. History of epilepsy
2. Sedatives
3. Muscle relaxants and epileptic prophylaxis within 24 hours

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic disorder of consciousness were enrolled in the Hangzhou Mingzhou Brain Rehabilitation Hospital, and healthy controls were all recorded by the First Affiliated Hospital of Zhejiang University.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Spectrum analysis of chronic disorders of consciousness | 6 months
  The EEG of 59 patients with disturbance of consciousness will be collected in resting state and listening to music, and the absolute power spectral density values (alpha,beta,theta,delta bands dB/Hz) will be calculated using spectral analysis.
Duration of each microstate | 6 months
  The investigators conducted resting state EEG recordings on 59 patients with consciousness disorders and 32 healthy controls. The investigators refined the microstate method to accurately estimate topographical differences. The calculations were performed for measures of duration (ms). The duration of each microstate were utilized to predict disease classification and prognosis evaluation for patients with disturbance of consciousness.
Occurrence of each microstate | 6 months
  The investigators conducted resting state EEG recordings on 59 patients with consciousness disorders and 32 healthy controls. The investigators refined the microstate analysis. The calculations were performed for measures of occurrence (times per minute). The occurrence of microstates were utilized to predict disease classification and prognosis evaluation for patients with disturbance of consciousness.
Global explained variance (GEV) of each microstate | 6 months
  The investigators conducted resting state EEG recordings on 59 patients with consciousness disorders and 32 healthy controls. The investigators refined the microstate analysis. The calculations were performed for measures of GEV (%). The GEV of microstates were utilized to predict disease classification and prognosis evaluation for patients with disturbance of consciousness.

SECONDARY OUTCOMES:
Coma Recovery Scale-Revised(CRS-R) | 30 minutes before samples collection
  The Coma Recovery Scale-Revised (CRS-R) score was utilized to measure the severity of the condition. It comprises 23 items arranged hierarchically into six subscales, including auditory, visual, motor, oromotor/verbal, communication, and arousal processes. Reflexive activity is represented by the lowest item on each subscale, while cognitively mediated behaviors are portrayed by the highest items. The scale ranges from 0 (indicating the lowest level of consciousness) to 23 (indicating the highest level of consciousness). Generally, a higher score suggests a better level of consciousness, while a lower score suggests a lower level of consciousness.
Glasgow Outcome Scale (GOS) | 6 months
  A GOS score ≥ 4 points is considered to indicate a good prognosis, while a GOS score < 4 points is considered to indicate a poor prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Benyuan Luo, Study Chair — Department of Neurology, First Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Yi Ling, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No